CLINICAL TRIAL: NCT00827567
Title: A Phase II Trial of RAD001 in Triple Negative Metastatic Breast Cancer
Brief Title: Trial of RAD001 in Triple Negative Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Allan Lipton, Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAD001JUS48T
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Results first posted 2012-04-20 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2013-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer; metastatic breast; triple negative; ER/PR negative; Her2 Neu negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD 001 (Experimental): RAD001-10 mg by mouth once everyday
  Interventions: Drug: RAD 001

INTERVENTIONS:
Drug: RAD 001 — RAD 001-10 mg by mouth once everyday
  Other Names: Everolimus

SUMMARY:
The hypothesis of this clinical research study is to discover if the study drug RAD001 can shrink or slow the growth of Estrogen Receptor/Progesterone Receptor (ER/PR) negative or Human Epidermal growth factor Receptor 2 (Her2 Neu) negative breast cancer. The safety of RAD001 will also be studied. Patients physical state, symptoms, changes in the size of the tumor, and laboratory findings obtained while on-study will help the research team decide if RAD001 is safe and effective.

DETAILED DESCRIPTION:
RAD001 is an orally administered cell cycle inhibitor with antitumor activity. RAD001, like Rapamycin, binds with high affinity to an intracellular immunophilin, FKBP12 and this complex specifically interacts with the mammalian target of rapamycin (mTOR) protein kinase, inhibiting downstream events such as the initiation of mRNA translation. RAD001 inhibits the growth of a wide range of histologically diverse tumor cells. RAD001 is being developed as a cytostatic agent to delay the time to tumor recurrence/progression or to increase survival in patients with various malignancies. The compound has good tolerability, a partially discovered mechanism of action. RAD001 has the ability to arrest cells in the G1 phase, and the ability to induce apoptosis. RAD001 is being investigated as an anticancer agent based on its potential to act directly on the tumor cells by inhibiting tumor cell growth and proliferation through possible inhibition of the PI3/AKT/MTOR pathway.

RAD001 was shown to have activity in human tumor cell lines originating from lung, breast, prostate, colon, kidney, melanoma and glioblastoma. RAD001 was also shown to have activity in human pancreatic neuroendocrine cells, where induction of apoptosis was reported, as well as in acute myeloid leukemia cells, adult T-cell leukemia cells, diffuse large B cell lymphoma cells, pancreatic tumor cells, ovarian cancer cells, and hepatocellular carcinoma cells.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Group (ECOG) performance status ≤ 2
* Age ≥ 18 years
* At least one measurable site of disease according to RECIST criteria that has not been previously irradiated. If the patient has had previous radiation to the marker lesion(s), there must be evidence of disease progression since the radiation
* Adequate bone marrow function as shown by: Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L, Platelets (PLT)≥ 100 x 109/L, Hemoglobin (HGB) ≥9 g/dL
* Adequate liver function as shown by:Serum bilirubin ≤ 1.5 x upper limits of normal (ULN), Prothrombin Time (INR) ≤ 1.3 (or ≤ 3 on anticoagulants), Liver function teats ≤ 2.5x ULN (≤ 5x ULN in patients with liver metastases)
* Adequate renal function: serum creatinine ≤ 1.5 x ULN
* Controlled diabetes as defined by fasting serum glucose ≤1.5 x ULN
* Fasting serum cholesterol ≤300 mg/dL or ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN.

Exclusion Criteria:

* Currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, antibody based therapy, etc.)
* Palliative radiation therapy only allowed to localized areas (ie: painful rib lesion), at the discretion of the PI and treating radiation oncologist
* Major surgery/significant traumatic injury within 4 weeks of start of study drug.
* Not recovered from the side effects of any major surgery (defined as requiring general anesthesia) to Grade I or patients that may require major surgery during the course of the study.
* Prior treatment with any investigational drug within the preceding 4 weeks
* Receiving chronic immunosuppressive agents, except corticosteroids with a daily dosage equivalent to prednisone ≤ 20 milligrams (mg). However, patients receiving corticosteroids must have been on a stable dosage regimen for a minimum of 4 weeks prior to the first treatment with RAD001. Topical or inhaled corticosteroids are allowed.
* May not receive immunization with attenuated live vaccines within one week of study entry or during study period.
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Other malignancies within the past 3 years, except for adequately treated carcinoma of the cervix and basal or squamous cell carcinomas of the skin.
* Severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as: Congestive heart failure: New York Heart Association Class III/IV, Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease.
* Impaired lung function (PFT screen at baseline) as defined as spirometry and DLCO that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air.
* Uncontrolled diabetes as defined by fasting serum glucose ≥1.5 x ULN. Glucose control should be achieved before starting a patient on RAD001.
* Active (acute or chronic) or uncontrolled severe infections
* Liver disease(cirrhosis, chronic active hepatitis or chronic persistent hepatitis)
* Known history of Human Immunodeficiency Virus (HIV) seropositivity
* Impairment of gastrointestinal function/disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Active, bleeding diathesis
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods.
* Prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus).
* Known hypersensitivity to RAD001 (everolimus) or other rapamycin drugs (sirolimus, temsirolimus) or to its excipients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Lipton, MD, Principal Investigator — Penn State Milton S. Hershey
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Atkins MB, Hidalgo M, Stadler WM, Logan TF, Dutcher JP, Hudes GR, Park Y, Liou SH, Marshall B, Boni JP, Dukart G, Sherman ML. Randomized phase II study of multiple dose levels of CCI-779, a novel mammalian target of rapamycin kinase inhibitor, in patients with advanced refractory renal cell carcinoma. J Clin Oncol. 2004 Mar 1;22(5):909-18. doi: 10.1200/JCO.2004.08.185. PMID 14990647
- [Background] Baselga, J. et al. Improved clinical and cell cycle response with an mTOR inhibitor, daily oral RAD001 (everolimus) plus letrozole versus placebo plus letrozole in a randomized phase II neoadjuvant trial in ER+ breast cancer. J Clin Oncol 26: 2008 (May 20 suppl; abstr 530)
- [Background] Bjornsti MA, Houghton PJ. The TOR pathway: a target for cancer therapy. Nat Rev Cancer. 2004 May;4(5):335-48. doi: 10.1038/nrc1362. No abstract available. PMID 15122205
- [Background] Bose S, Chandran S, Mirocha JM, Bose N. The Akt pathway in human breast cancer: a tissue-array-based analysis. Mod Pathol. 2006 Feb;19(2):238-45. doi: 10.1038/modpathol.3800525. PMID 16341149
- [Background] Boulay A, Lane HA. The mammalian target of rapamycin kinase and tumor growth inhibition. Recent Results Cancer Res. 2007;172:99-124. doi: 10.1007/978-3-540-31209-3_7. No abstract available. PMID 17607938
- [Background] Eisen HJ, Tuzcu EM, Dorent R, Kobashigawa J, Mancini D, Valantine-von Kaeppler HA, Starling RC, Sorensen K, Hummel M, Lind JM, Abeywickrama KH, Bernhardt P; RAD B253 Study Group. Everolimus for the prevention of allograft rejection and vasculopathy in cardiac-transplant recipients. N Engl J Med. 2003 Aug 28;349(9):847-58. doi: 10.1056/NEJMoa022171. PMID 12944570
- [Background] Haritunians T, Mori A, O'Kelly J, Luong QT, Giles FJ, Koeffler HP. Antiproliferative activity of RAD001 (everolimus) as a single agent and combined with other agents in mantle cell lymphoma. Leukemia. 2007 Feb;21(2):333-9. doi: 10.1038/sj.leu.2404471. Epub 2006 Nov 30. PMID 17136116
- [Background] Ingelman-Sundberg M. Human drug metabolising cytochrome P450 enzymes: properties and polymorphisms. Naunyn Schmiedebergs Arch Pharmacol. 2004 Jan;369(1):89-104. doi: 10.1007/s00210-003-0819-z. Epub 2003 Oct 22. PMID 14574440
- [Background] Ikezoe T, Nishioka C, Bandobashi K, Yang Y, Kuwayama Y, Adachi Y, Takeuchi T, Koeffler HP, Taguchi H. Longitudinal inhibition of PI3K/Akt/mTOR signaling by LY294002 and rapamycin induces growth arrest of adult T-cell leukemia cells. Leuk Res. 2007 May;31(5):673-82. doi: 10.1016/j.leukres.2006.08.001. Epub 2006 Sep 27. PMID 17007924
- [Background] Jerusalem G.H et al. Multicenter phase I clinical trial of daily and weekly RAD001 in combination with vinorelbine and trastuzumab in patients with HER2-overexpressing metastatic breast cancer with prior resistance to trastuzumab. J Clin Oncol 26: 2008 (May 20 suppl; abstr 1057)
- [Background] Tanaka C, O'Reilly T, Kovarik JM, Shand N, Hazell K, Judson I, Raymond E, Zumstein-Mecker S, Stephan C, Boulay A, Hattenberger M, Thomas G, Lane HA. Identifying optimal biologic doses of everolimus (RAD001) in patients with cancer based on the modeling of preclinical and clinical pharmacokinetic and pharmacodynamic data. J Clin Oncol. 2008 Apr 1;26(10):1596-602. doi: 10.1200/JCO.2007.14.1127. Epub 2008 Mar 10. PMID 18332467
- [Background] Mabuchi S, Altomare DA, Cheung M, Zhang L, Poulikakos PI, Hensley HH, Schilder RJ, Ozols RF, Testa JR. RAD001 inhibits human ovarian cancer cell proliferation, enhances cisplatin-induced apoptosis, and prolongs survival in an ovarian cancer model. Clin Cancer Res. 2007 Jul 15;13(14):4261-70. doi: 10.1158/1078-0432.CCR-06-2770. PMID 17634556
- [Background] Manning BD, Cantley LC. AKT/PKB signaling: navigating downstream. Cell. 2007 Jun 29;129(7):1261-74. doi: 10.1016/j.cell.2007.06.009. PMID 17604717
- [Background] Mondesire WH, Jian W, Zhang H, Ensor J, Hung MC, Mills GB, Meric-Bernstam F. Targeting mammalian target of rapamycin synergistically enhances chemotherapy-induced cytotoxicity in breast cancer cells. Clin Cancer Res. 2004 Oct 15;10(20):7031-42. doi: 10.1158/1078-0432.CCR-04-0361. PMID 15501983
- [Background] Sieghart W, Fuereder T, Schmid K, Cejka D, Werzowa J, Wrba F, Wang X, Gruber D, Rasoul-Rockenschaub S, Peck-Radosavljevic M, Wacheck V. Mammalian target of rapamycin pathway activity in hepatocellular carcinomas of patients undergoing liver transplantation. Transplantation. 2007 Feb 27;83(4):425-32. doi: 10.1097/01.tp.0000252780.42104.95. PMID 17318075

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period 4/13/2009 through 2/25/2011. Protocol dated 3/6/2009 & consent dated 4/8/2009 for the 4/13/2009 approval.Patients were seen at Penn State Cancer Institute Outpatient Unit.
Pre-assignment Details: Two of the patients that were screen failures had cholesterol levels higher than inclusion criteria as this drug may increase cholesterol levels they were not eligible.
Period: Overall Study
Arm/Group | RAD 001
Started | 4
Completed | 0 (2 screen failures, 4 withdrew from study to go on to other therapies)
Not Completed | 4
Not completed — Progression of Disease/Screen Failure | 4

BASELINE CHARACTERISTICS:
Arm/Group | RAD 001
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (7.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression(TTP)
Description: Progression is defined by RESIST criteria as any new lesion or the sum of target lesions increasing by 20% over baseline
Time Frame: Each patient assessed at 8 weeks from start of study drug
Arm/Group | RAD 001
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Weekly for 4 weeks, then monthly until disease progression
Arm/Group | RAD 001
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD 001 (N=4)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes